CLINICAL TRIAL: NCT03549234
Title: A Randomized, Subject-Masked, Active-Controlled, Parallel-Arm Clinical Trial Comparing Erector Spinae and Paravertebral Nerve Blocks
Brief Title: Erector Spinae Versus Paravertebral Nerve Blocks for Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Erector Spinae vs PVB
Record Dates: First submitted 2018-04-24; First posted 2018-06-07 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Breast Surgery
Keywords: Regional anesthesia; Paravertebral; Erector spinae; Nerve block
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erector Spinae (single injection) (Experimental)
  Interventions: Drug: Erector Spinae (single injection)
- Paravertebral (single injection) (Active Comparator)
  Interventions: Drug: Paravertebral (single injection)

INTERVENTIONS:
Drug: Erector Spinae (single injection) — Ropivacaine 0.5% (with epinephrine 1:200,000-400,000) will be administered via the needle into the target plane.
  Arms: Erector Spinae (single injection)
Drug: Paravertebral (single injection) — Ropivacaine 0.5% (with epinephrine 1:200,000-400,000) will be administered via the needle into the target plane.
  Arms: Paravertebral (single injection)

SUMMARY:
Following painful surgical procedures of the breast, postoperative analgesia is often provided with a paravertebral nerve block (PVB). For intense, but shorter-duration acute pain, a single-injection of local anesthetic is used with a duration of approximately 12 hours. The PVB has several limitations: it can decrease blood pressure, and very rare-but serious-complications have occurred, including neuraxial injection, neuraxial hematoma, and pleural puncture. An alternative block has been described: the erector spinae plane block. The theoretical benefits include ease of administration since it is a plane superficial to the PVB and therefore easier to identify and target with ultrasound (therefore increasing success rate); and an increased safety margin: there are few anatomic structures in the immediate area which could be injured with the needle; and, the target plane is much further from the intrathecal/epidural space relative to the PVB. Lastly, the plane may be easier to catheterize for continuous peripheral nerve blocks relative to the relatively-small volume PVB.

There are therefore multiple theoretical reasons to prefer the erector spinae plane block. Unfortunately, it remains unknown if the analgesia provided by this new technique is comparable to that provided with the PVB. The investigators therefore propose to compare these two techniques with a randomized, subject-masked, active-controlled, parallel-arm, human subjects clinical trial.

DETAILED DESCRIPTION:
This investigation will be a randomized, subject-masked, active-controlled parallel-arm, human subjects clinical trial. Of note, the investigators will be using standard-of-care local anesthetic under an FDA-approved purpose and do not plan to research a possible change of indication or use of these medications as part of this research project. The treatments in both groups are currently used at the study institution and there is true clinical equipoise at this time. The only difference in treatment between subjects who enroll versus those not enrolled in this study will be those who enroll will have the decision between which anatomic block location determined randomly, as opposed to the physician simply choosing him/herself.

Enrollment. Consenting adults undergoing breast surgery with a planned single-injection regional analgesic will be offered enrollment. Patients undergoing breast surgery with a planned perineural catheter regional analgesic will be excluded. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current University of California San Diego (UCSD) Institutional Review Board (IRB)-approved Informed Consent Form (ICF). Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status. Inclusion and exclusion criteria are listed in another section.

Preoperative Procedures. Following written, informed consent, the investigators will collect baseline anthropomorphic information (e.g., age, sex, height, and weight). All subjects will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and placed in the sitting position. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. Both possible block locations will be viewed with ultrasound. If one or both of the locations is unacceptable for block placement in the clinician's opinion, the subject will not be randomized and will not proceed further with the study.

Subjects will then be randomized using a computer-generated list and opaque, sealed envelopes to one of two treatment groups: (blocks of 4, stratified for unilateral vs. bilateral surgery): (1) erector spinae plane or (2) paravertebral block. All blocks will be placed by a regional anesthesia fellow or resident under the direct supervision and guidance of a regional anesthesia attending (or by the attending him/herself).

The area of needle insertion will be cleaned with chlorhexidine gluconate and isopropyl alcohol. All blocks will be placed using standard UCSD ultrasound-guided techniques.

Ropivacaine 0.5% (with epinephrine 1:200,000-400,000) will be administered via the needle into the target plane. For erector spinae plane blocks, this will be at the T3 level for surgery involving the axilla and the T4 level for surgery not involving the axilla (20 mL of local anesthetic for unilateral surgery; 16 mL of local anesthetic each side for bilateral surgery). For PVBs without axillary work, this will be at the T3 and T5 levels. For PVBs with axillary work, this will be at the T2 and T4 levels. For unilateral PVBs, 10 mL of local anesthetic will be injected per level. For bilateral PVBs, 8 mL of local anesthetic will be injected per level.

Single-injection blocks will be considered successful if, within 30 minutes, the subject experiences decreased sensation to cold temperature with an alcohol pad over the approximate level of the ipsilateral 4th thoracic dermatome. Misplaced blocks will be replaced successfully, or the patient excluded from further study participation. For subjects undergoing bilateral surgical procedures, a block using the same protocol will be administered on the contralateral side.

Intraoperatively, all subjects will receive a general anesthetic using inhaled and intravenous anesthetic and oxygen. Intravenous fentanyl will be administered for cardiovascular responsiveness to noxious stimuli at the discretion of the anesthesia provider.

Postop: Subjects will be discharged with a prescription for oxycodone 5 mg tablets for supplementary analgesia and instructed to record the time at which subjects take their first opioid tablet as well as the time at which subjects believe the block starts to wear off.

Outcome measurements (end points). Pain scores will be recorded using the Numeric Rating Scale (NRS). Within the recovery room, pain scores, opioid requirements, and antiemetic administration will be recorded by nursing staff masked to treatment group. The morning following surgery, all subjects will be contacted by phone or in person [if hospitalized] to record lowest, average, highest, and current pain scores; sleep disturbances, and nausea using a 0-10 Likert scale (0 = no nausea; 10 = vomiting). For outpatients, opioid requirements will be recorded while inpatients will have opioid requirements extracted from the electronic medical record. In addition, the investigators will extract antiemetic use from the electronic record. The investigators will collect the times at which subjects felt their block resolve and subjects consumed their first opioid analgesic pills following recovery room discharge.

Hypothesis 1: Following breast surgery, analgesia will be non-inferior in the recovery room with an erector spinae plane block compared with a paravertebral block as measured with the Numeric Rating Scale.

Hypothesis 2: For breast surgery, opioid consumption will be non-inferior in the operating and recovery rooms with an erector spinae plane block compared with a paravertebral block (primary: cumulative intravenous morphine equivalents).

Primary end point: In order to claim that erector spinae plane blocks are non-inferior to paravertebral blocks, both Hypotheses 1 and 2 must be at least non-inferior.

Statistical methods. Descriptive statistics will be provided by arm and in aggregate. Baseline characteristics of arms will be compared using the Wilcoxon-Mann-Whitney and Fisher's Exact tests. Key characteristics that are significantly different (p<0.05) will be included as covariates in the analysis models.

Primary aim. The investigators will test the noninferiority of the erector spinae nerve block compared to the paravertebral nerve block. The 95% confidence interval (CI) associated with the Wilcoxon-Mann-Whitney test will be derived for the group difference (paravertebral minus erector spinae) in median pain scores within the recovery room. If the lower limit of the 95% CI is greater than -1.25, the investigators will conclude noninferiority. If there are significant differences between the groups in any key characteristics, these characteristics will be included as covariates in a linear model. The same noninferiority margin (-1.25) will be applied to the 95% CI for the covariate adjusted group difference in mean pain derived from the linear model.

The noninferiority of the erector spinae nerve block with regard to total opioid consumption within the operating and recovery rooms will be tested in the same manner as pain, i.e. comparing the limits of a 95% CI associated with the Wilcoxon-Mann-Whitney test to a predefined noninferiority margin (in this case 2 mg). Covariate adjusted linear models will again be applied in the event that key characteristics are significantly different between the groups.

Sample size justification. Power for the Wilcoxon-Mann-Whitney derived noninferiority testing is based on 10,000 simulated trials. The investigators simulated pain scores from a discrete distribution with median (interquartile range) 3 (2-5) [Kairaluoma, 2004]. Between the quartiles, the probability of each score was assumed constant. The distribution for each group was assumed to be the same. The sample size of n=50 per group provides 82% power to detect noninferiority in pain with a margin of 1.25. Similarly, opioid consumption was assumed to follow a truncated normal distribution with mean 2.5 mg and standard deviation 2 mg, and minimum value 0 mg. The sample size of n = 50 per group provides at least 95% power to detect noninferiority with margin 2 mg. Therefore, the investigators will enroll 50 subjects for each of two treatments with a total enrollment of 100 subjects. To allow for dropouts, the investigators will request a maximum enrollment of 120 subjects. Noninferiority in pain is tested first, and if significant, noninferiority in opioid consumption is tested. Under this hierarchical testing framework, no adjustment in alpha is necessary to control Type 1 error [Mascha, et al 2012].

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral or bilateral breast surgery with at least moderate postoperative pain anticipated
* analgesic plan includes a single-injection peripheral nerve block(s)
* age 18 years or older.

Exclusion Criteria:

* morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2)
* renal insufficiency (preoperative creatinine > 1.5 mg/dL)
* chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* history of opioid abuse
* any comorbidity which results in moderate or severe functional limitation
* inability to communicate with the investigators or hospital staff
* pregnancy
* planned regional analgesic with perineural catheter placement
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD MS, Principal Investigator — Professor in Residence
Locations (1):
- UCSD Medical Center (Hillcrest and Thornton), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naja Z, Lonnqvist PA. Somatic paravertebral nerve blockade. Incidence of failed block and complications. Anaesthesia. 2001 Dec;56(12):1184-8. doi: 10.1046/j.1365-2044.2001.02084-2.x. PMID 11736777
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] Ilfeld BM, Madison SJ, Suresh PJ, Sandhu NS, Kormylo NJ, Malhotra N, Loland VJ, Wallace MS, Proudfoot JA, Morgan AC, Wen CH, Wallace AM. Treatment of postmastectomy pain with ambulatory continuous paravertebral nerve blocks: a randomized, triple-masked, placebo-controlled study. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):89-96. doi: 10.1097/AAP.0000000000000035. PMID 24448512
- [Background] Finneran JJ 4th, Gabriel RA, Khatibi B. Erector Spinae Plane Blocks Provide Analgesia for Breast and Axillary Surgery: A Series of 3 Cases. Reg Anesth Pain Med. 2018 Jan;43(1):101-102. doi: 10.1097/AAP.0000000000000695. No abstract available. PMID 29261601
- [Background] Kairaluoma PM, Bachmann MS, Korpinen AK, Rosenberg PH, Pere PJ. Single-injection paravertebral block before general anesthesia enhances analgesia after breast cancer surgery with and without associated lymph node biopsy. Anesth Analg. 2004 Dec;99(6):1837-1843. doi: 10.1213/01.ANE.0000136775.15566.87. PMID 15562083
- [Background] Mascha EJ, Turan A. Joint hypothesis testing and gatekeeping procedures for studies with multiple endpoints. Anesth Analg. 2012 Jun;114(6):1304-17. doi: 10.1213/ANE.0b013e3182504435. Epub 2012 May 3. PMID 22556210
- [Derived] Swisher MW, Wallace AM, Sztain JF, Said ET, Khatibi B, Abanobi M, Finneran Iv JJ, Gabriel RA, Abramson W, Blair SL, Hosseini A, Dobke MK, Donohue MC, Ilfeld BM. Erector spinae plane versus paravertebral nerve blocks for postoperative analgesia after breast surgery: a randomized clinical trial. Reg Anesth Pain Med. 2020 Apr;45(4):260-266. doi: 10.1136/rapm-2019-101013. Epub 2020 Jan 21. PMID 31969443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection) | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 33 | 72
  >=65 years | 11 | 17 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.5 [48 to 63.8] | 54.5 [44 to 67.8] | 54.5 [47 to 65.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale Pain Scores
Description: Range scale minimum 0, maximum 10. Lower pain scores are considered a better outcome, higher pain scores are considered a worse outcome.
Time Frame: 1 day (PACU pain scores)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 50 | 50
score on a scale | 3.0 [0.25 to 5] | 0 [0 to 3.13]
Statistical Analysis 1: Comparison: Erector Spinae (Single Injection) vs Paravertebral (Single Injection); We hypothesized that 1) analgesia would be noninferior in the recovery room as measured on a Numeric Rating Scale with ESPB (erector spinae plane block), and 2) opioid consumption would be noninferior in the operating and recovery rooms with ESPB. We simulated pain scores from a discrete distribution with median (interquartile range) 2 (0-3). The sample size of 50 per group provided 81% power to detect noninferiority in pain; Test type: Non-Inferiority — We tested the noninferiority of ESPB compared to PVB (paravertebral block) using the 95% confidence interval (CI) associated with the Wilcoxon-Mann-Whitney Exact test. If the lower limit of the 95% CI for median "average" recovery room pain scores was greater than -1.25 (based on PVB minus ESPB), we concluded noninferiority. The noninferiority of ESPBs with regard to opioid consumption was similarly tested with a predefined noninferiority margin of 2 mg intravenous morphine equivalents; p = 0.0011, Wilcoxon (Mann-Whitney)

2. Primary Outcome: OR and PACU Opioid Consumption
Description: This outcome measure reflects the total amount of opioid administered in the operating room and recovery room perioperatively. Specific time points are not applicable since operating room and recovery room times differ among subjects.
Time Frame: up to 1 day, in the OR and PACU
Measure: Median (Inter-Quartile Range); unit: morphine equivalents
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 50 | 50
morphine equivalents | 2.0 [1.14 to 4.52] | 1.4 [1.00 to 2.07]
Statistical Analysis 1: Comparison: Erector Spinae (Single Injection) vs Paravertebral (Single Injection); Test type: Non-Inferiority — We tested the noninferiority of ESPB compared to PVB using the 95% confidence interval (CI) associated with the Wilcoxon-Mann-Whitney Exact test. If the lower limit of the 95% CI for median "average" recovery room pain scores was greater than -1.25 (based on PVB minus ESPB), we concluded noninferiority. The noninferiority of ESPBs with regard to opioid consumption was similarly tested with a predefined noninferiority margin of 2 mg intravenous morphine equivalents; p = 0.0043, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Nausea and Vomiting
Description: Nausea and vomiting was recorded using a 0-10 Likert scale (0 = no nausea; 10 = vomiting) on postoperative day 1. Higher scores represent a worse outcome.
Time Frame: postoperative day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 50 | 50
score on a scale | 0 [0 to 0] | 0 [0 to 0]

4. Other Pre Specified Outcome: Sleep Disturbances
Time Frame: postoperative day 1
Measure: Median (Inter-Quartile Range); unit: awakenings
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 50 | 50
awakenings | 0 [0 to 0] | 0 [0 to 1]

5. Other Pre Specified Outcome: Time of Block Resolution
Description: This was recorded as the time at which a participant subjectively noticed that the nerve block was wearing off and sensation was returning.
Time Frame: postoperative day 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 50 | 50
hours | 17.7 [9.66 to 20.07] | 16.0 [11.88 to 19.93]

6. Other Pre Specified Outcome: Opioid Consumption
Description: Number of oxycodone tablets (in mg) taken by the participant after discharge from the recovery room was recorded during follow-up on postoperative day 1.
Time Frame: postoperative day 1
Measure: Median (Inter-Quartile Range); unit: mg oxycodone
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
Number analyzed (Participants) | 50 | 50
mg oxycodone | 5 [0 to 10] | 10 [0 to 15]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Erector Spinae (Single Injection) | Paravertebral (Single Injection)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03549234/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03549234/Prot_SAP_002.pdf